CLINICAL TRIAL: NCT00392678
Title: Targeting Inflammation in Type 2 Diabetes: Clinical Trial Using Salsalate
Brief Title: Targeting INflammation Using SALsalate in Type 2 Diabetes (TINSAL-T2D)
Acronym: TINSAL-T2D
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS 06-20, NIH U01 DK74556; U01DK074556 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-07-26 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Inflammation; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Obesity; Metabolic Syndrome | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo, appearance matched to active drug
  Interventions: Drug: Placebo
- 3 gram (Active Comparator): Salsalate 3.0 grams daily, divided
  Interventions: Drug: Salsalate
- 3.5 gram (Active Comparator): Salsalate 3.5 g daily, divided
  Interventions: Drug: Salsalate
- 4 gram (Active Comparator): Salsalate 4.0 g daily, divided
  Interventions: Drug: Salsalate

INTERVENTIONS:
Drug: Salsalate — Placebo and Salsalate 3.0 g/d; 3.5 g/d; 4.0 g/d orally, divided
  Other Names: Disalcid; Salicylsalicylic acid
  Arms: 3 gram; 3.5 gram; 4 gram
Drug: Placebo — Placebo to Salsalate
  Other Names: Placebo to Salsalate
  Arms: Placebo

SUMMARY:
Growing evidence over recent years supports a potential role for low grade chronic inflammation in the pathogenesis of insulin resistance and type 2 diabetes. In this study we will determine whether salsalate, a member of the commonly used Non-Steroidal Anti-Inflammatory Drug (NSAID) class, is effective in lowering sugars in patients with type 2 diabetes. The study will determine whether salicylates represent a new pharmacological option for diabetes management. The study is conducted in two stages. The first stage is a dose ranging study, administering salsalate compared to placebo over three months. The primary objective of Stage 2 of the study is to evaluate the effects of salsalate on blood sugar control in diabetes; the tolerability of salsalate use in patients with type 2 diabetes (T2D); and the effects of salsalate on measures of inflammation, the metabolic syndrome, and cardiac risk.

The second stage is a second trial and posted under alternate registration.

DETAILED DESCRIPTION:
The primary objective of the first stage of the TINSAL-T2D trial is to select a dose of salsalate that is both well-tolerated and demonstrates a trend toward improvement in glycemic control. The trial is a multicenter, single mask lead-in, double masked placebo controlled dose ranging study, comparing salsalte to placebo over 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes on diet and exercise therapy or monotherapy with metformin, insulin secretagogue, or alpha-glucosidase inhibitors, or a low-dose combination of these at ≤ 50% maximal dose (see Appendix). Dosing is stable for 8 weeks prior to randomization.
2. FPG ≤ 225 mg/dL and HbA1c>7% and ≤9.5% at screening
3. Age ≥18 and <75
4. Women of childbearing potential agree to use an appropriate contraceptive method (hormonal, IUD, or diaphragm)

Exclusion Criteria:

1. Type 1 diabetes and/or history of ketoacidosis determined by medical history
2. History of severe diabetic neuropathy including autonomic neuropathy, gastroparesis or lower limb ulceration or amputation
3. History of long-term therapy with insulin (>30 days) within the last year
4. Therapy with rosiglitazone (Avandia) or pioglitazone (Actos), or extendin-4 (Byetta), alone or in combination in the previous 6 months
5. Pregnancy or lactation
6. Patients requiring corticosteroids within 3 months or recurrent continuous oral corticosteroid treatment (more than 2 weeks)
7. Use of weight loss drugs [e.g., Xenical (orlistat), Meridia (sibutramine), Acutrim (phenylpropanol-amine), or similar over-the-counter medications] within 3 months of screening or intentional weight loss of ≥ 10 lbs in the previous 6 months
8. Surgery within 30 days prior to screening
9. Serum creatinine >1.4 for women and >1.5 for men or eGFR <60 [possible chronic kidney disease stage 3 or greater calculated using the Modification of Diet in Renal Disease (MDRD) equation.
10. History of chronic liver disease including hepatitis B or C
11. History of peptic ulcer or endoscopy demonstrated gastritis
12. History of acquired immune deficiency syndrome or human immunodeficiency virus (HIV)
13. History of malignancy, except participants who have been disease-free for greater than 10 years, or whose only malignancy has been basal or squamous cell skin carcinoma
14. New York Heart Association Class III or IV cardiac status or hospitalization for congestive heart failure
15. History of unstable angina, myocardial infarction, cerebrovascular accident, transient ischemic attack or any revascularization within 6 months
16. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg on three or more assessments on more than one day)
17. History of drug or alcohol abuse, or current weekly alcohol consumption >10 units/week (1 unit = 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 ounce of alcohol)
18. Hemoglobin <12 g/dL (males), <10 g/dL (females) at screening
19. Platelets <100,000 cu mm at screening.
20. AST (SGOT) >2.50 x ULN or ALT (SGPT) >2.50 x ULN at screening
21. Total Bilirubin >1.50 x ULN at screening
22. Triglycerides (TG) >500 mg/dL at screening
23. Poor mental function or any other reason to expect patient difficulty in complying with the requirements of the study
24. Previous allergy to aspirin
25. Chronic or continuous use (daily for more than 7 days) of nonsteroidal anti-inflammatory drugs within the preceding 2 months
26. Use of warfarin (Coumadin), clopidogrel (Plavix) or other anticoagulants
27. Use of probenecid (Benemid, Probalan), sulfinpyrazone (Anturane) or other uricosuric agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Sheolson, MD, PhD, Principal Investigator — Joslin Diabetes Center; Allison B. Goldfine, MD, Study Director — Joslin Diabetes Center; Vivian Fonseca, MD, Study Director — Tulane University; Kathleen Jablonski, PhD, Study Director — George Washington University; Myrlene Staten, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (16):
- United States (16):
  - Chapel Medical Group, New Haven, Connecticut
  - MedStar Research Institute, Washington D.C., District of Columbia
  - Endocrine Clinical Research, Winter Park, Florida
  - Kaiser Permanente, Atlanta, Georgia
  - Emory School of Medicine, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Kaleida Health Center, Buffalo, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Chen YD, Tipton L, Staten MA, Shoelson SE; Targeting Inflammation Using Salsalate in Type 2 Diabetes Study Team. Salicylate (salsalate) in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2013 Jul 2;159(1):1-12. doi: 10.7326/0003-4819-159-1-201307020-00003. PMID 23817699
- [Result] Goldfine AB, Fonseca V, Jablonski KA, Pyle L, Staten MA, Shoelson SE; TINSAL-T2D (Targeting Inflammation Using Salsalate in Type 2 Diabetes) Study Team. The effects of salsalate on glycemic control in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2010 Mar 16;152(6):346-57. doi: 10.7326/0003-4819-152-6-201003160-00004. PMID 20231565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 private practices and 14 universities. First patient recruited February 2007; last patient end of study visit, May 2008
Pre-assignment Details: Screening, followed by 4-week single mask placebo lead-in. 277 participants signed screening consent. Some participants were ineligible, some withdrew consent, and some had treatment side effects during placebo lead-in.
Groups:
- 3 Gram: Salsalate 3.0 g daily, divided
- Placebo: Matched by appearance to active drug
Period: Overall Study
Arm/Group | 3 Gram | 3.5 Gram | 4 Gram | Placebo
Started | 27 | 27 | 27 | 27
Completed | 27 | 26 | 25 | 26
Not Completed | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: matched to active drug
- Total: Total of all reporting groups
Arm/Group | 3 Gram | 3.5 Gram | 4 Gram | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 24 | 22 | 91
  >=65 years | 4 | 5 | 3 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (9.4) | 56.7 (9.8) | 55.0 (10.2) | 55.9 (8.2) | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 11 | 12 | 45
  Male | 14 | 18 | 16 | 15 | 63
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 27 | 27 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c Baseline to End of Trial in TINSAL-T2D Stage 1
Description: The primary outcome for the TINSAL-T2D study is change in HbA1c level from baseline to week 14 (stage 1) in the intent-to-treat (ITT) population with last observation carried forward.
Time Frame: 14 week
Measure: Mean (95% Confidence Interval); unit: % (units of HbA1c)
Groups:
- 3.0 g/d: Salsalate 3.0 g/d, divided
- 3.5 g/d: Salsalate 3.5 g/d, divided
- 4.0 g/d: Salsalate 4.0 g/d, divided
- Placebo: Placebo matched to active drug
Arm/Group | 3.0 g/d | 3.5 g/d | 4.0 g/d | Placebo
Number analyzed (Participants) | 27 | 26 | 25 | 26
% (units of HbA1c) | -0.36 [-0.55 to -0.17] | -0.34 [-0.54 to -0.15] | -0.49 [-0.69 to -0.30] | -0.01 [-0.20 to 0.19]
Statistical Analysis 1: Comparison: 3.0 g/d vs 3.5 g/d vs 4.0 g/d vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Change in HbA1c
Description: Change from baseline to either 14 or 26 weeks, or last HbA1c measurement prior to rescue therapy
Time Frame: 14 week
Measure: Mean (95% Confidence Interval); unit: % HbA1c
Groups:
- Salsalate 3.0 g/d: Salsalate 3.0 g/d, divided
- Salsalate 3.5 g/d: Salsalate 3.5 g/d, divided
- Salsalate 4.0 g/d: Salsalate 4.0 g/d, divided
Arm/Group | Placebo | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d
Number analyzed (Participants) | 26 | 27 | 26 | 25
% HbA1c | 0 [-0.2 to 0.2] | -0.4 [-0.6 to -0.2] | -0.3 [-0.5 to -0.2] | -0.5 [-0.7 to -0.3]

3. Secondary Outcome: Change From Baseline and Trends in Fasting Glucose Over Time
Time Frame: 14 week
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Placebo | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d
Number analyzed (Participants) | 26 | 27 | 26 | 25
mg/dl | 13 [2 to 24] | -19 [-30 to -8] | -14 [-25 to -3] | -15 [-26 to -4]

4. Secondary Outcome: Change in Lipids
Description: Change in lipids (low-density lipoprotein cholesterol [LDL-C], non-high-density lipoprotein cholesterol [non-HDL-C], triglycerides [TG], total cholesterol [TC], high-density lipoprotein cholesterol [HDL C], TC/HDL-C ratio, and LDL-C/HDL-C ratio)
  LDL-C/HDL-C ratio not calculated
Time Frame: 14 week
Measure: Mean (95% Confidence Interval); unit: mg/dl
Groups:
- Placebo: Placebo matched to active
Arm/Group | Placebo | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d
Number analyzed (Participants) | 26 | 27 | 26 | 27
mg/dl
  Cholesterol | 0 [-7 to 8] | 8 [1 to 16] | -1 [-9 to 7] | 6 [-1 to 14]
  HDL | 0 [-2 to 1] | 3 [1 to 4] | 1 [-1 to 3] | 2 [0 to 4]
  LDL | 0 [-7 to 6] | 15 [9 to 22] | 3 [-3 to 10] | 8 [2 to 15]
  TG | 15 [-6 to 36] | -34 [-55 to -13] | -22 [-43 to 0] | -16 [-38 to 5]
  Total to HDL ratio | 0 [-0.2 to 0.3] | 0.1 [-0.1 to 0.4] | -0.1 [-0.3 to 0.2] | 0.2 [-0.1 to 0.4]

5. Secondary Outcome: Change From Baseline in 14-week Insulin, C-peptide, Homeostasis Model [HOMA] Index
Description: HOMA-IR was not calcuated due to potential confounding effect of salicylates to inhibit insulin clearance. Change in insulin from Baseline to Week 14 in data table below.
Time Frame: Baseline, week 14
Measure: Median (Inter-Quartile Range); unit: pmol/l
Arm/Group | Placebo | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d
Number analyzed (Participants) | 26 | 27 | 26 | 25
pmol/l | -3.0 [-39 to 33] | 15 [12 to 42] | 7.6 [-21.4 to 36.6] | 27 [-31 to 85]

6. Secondary Outcome: Safety and Tolerability
Description: See adverse event module for details. Safety and tolerability of salsalate compared to placebo as assessed by adverse events.
Time Frame: 14 weeks
Measure: Number; unit: participants
Arm/Group | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d | Placebo
Number analyzed (Participants) | 27 | 27 | 27 | 27
participants | 17 | 16 | 16 | 14

7. Secondary Outcome: Change in Insulin, C-peptide, Homeostasis Model [HOMA] Index
Description: HOMA-IR was not calcuated due to potential confounding effect of salicylates to inhibit insulin clearance. Change in C-peptide from Baseline to Week 14 is in the data table below
Time Frame: Baseline, week 14
Measure: Mean (95% Confidence Interval); unit: C-peptide in nmol/l
Arm/Group | Placebo | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d
Number analyzed (Participants) | 26 | 27 | 26 | 25
C-peptide in nmol/l | 0.10 [0 to 0.2] | -0.07 [-0.17 to 0.01] | -0.03 [-0.13 to 0.10] | 0.03 [-0.07 to 0.13]

ADVERSE EVENTS:
Time Frame: Screening, 4 week placebo run in, 14 week treatment.
Description: AE/SAE use standard FDA definition.
Groups:
- Salsalate 3.0 g/d: Active: Salsalate 3.0 g/d
- Salsalate 3.5 g/d: Active: Salsalate 3.5 g/d
- Salsalate 4.0 g/d: Active: Salsalate 4.0 g/d
- Placebo: Identical Placebo
Arm/Group | Salsalate 3.0 g/d | Salsalate 3.5 g/d | Salsalate 4.0 g/d | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27 | 2/27 | 0/27 | 1/27
Other Adverse Events (participants affected / at risk) | 27/27 | 27/27 | 27/27 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate 3.0 g/d (N=27) | Salsalate 3.5 g/d (N=27) | Salsalate 4.0 g/d (N=27) | Placebo (N=27)
Acute Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for Acute Cholecystitis, laparoscopic cholecystectomy performed.
Cervical Disc Herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — 1. Hospitalization for Cervical Disc Herniation.
Congestive Heart Failure with Diastolic Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hospitalization for Congestive Heart Failure with Diastolic Dysfunction.
Lumbar laminectomy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for Lumbar laminectomy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate 3.0 g/d (N=27) | Salsalate 3.5 g/d (N=27) | Salsalate 4.0 g/d (N=27) | Placebo (N=27)
Cardiorespiratory (Cardiac disorders) | 4 (5) | 1 (1) | 3 (5) | 3 (7) — Includes palpitations, chest pain or discomfort, and swelling of legs or feet
Neurologic (Nervous system disorders) | 7 (9) | 10 (13) | 8 (8) | 7 (7) — Includes blurry vision, dots or flashes in vision, tinnitus, and numbness or tingling.
Gastrointestinal (Gastrointestinal disorders) | 11 (13) | 8 (8) | 8 (8) | 2 (3) — incudes heartburn, nausea, vomiting, diarrhea
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (5) | 3 (3) | 7 (9) — Includes stiffness, muscle or joint pain, arthritis, backache.
General (General disorders) | 7 (8) | 4 (4) | 2 (2) | 4 (4) — Includes fainting, dizziness, weakness or fatigue.
Hypoglycemia (Endocrine disorders) | 5 (63) | 6 (46) | 6 (7) | 2 (2)
Hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No